CLINICAL TRIAL: NCT02446795
Title: Isoquercetin as an Adjunct Therapy in Patients With Kidney Cancer Receiving First-line Sunitinib: a Phase I/II Trial
Acronym: QUASAR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry); Quercegen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QUASAR - 2014-001; 2015-000194-12 (EudraCT Number)
Record Dates: First submitted 2015-05-06; First posted 2015-05-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
Keywords: Renal cell carcinoma; Isoquercetin; kidney cancer; sunitinib; fatigue
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Fatigue | interventions — Sunitinib; isoquercitrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm (Experimental): Phase I Sunitinib: 50mg once daily orally schedule treatment according to Investigator's choice Isoquercetin: 225mg twice a day (at 08 a.m. and at 4 p.m). Phase II Sunitinib: 50mg once daily orally schedule treatment according to Investigator's choice Isoquercetin: 450 mg twice a day (at 08 a.m. and at 4 p.m).
  Interventions: Drug: Sunitinib; Drug: Isoquercetin
- Placebo Arm (Placebo Comparator): Phase I Sunitinib: 50mg once daily orally schedule treatment according to Investigator's choice Placebo: 225mg twice a day (at 08 a.m. and at 4 p.m). Phase II Sunitinib: 50mg once daily orally schedule treatment according to Investigator's choice Placebo: 450 mg twice a day (at 08 a.m. and at 4 p.m).
  Interventions: Drug: Sunitinib; Drug: Placebo

INTERVENTIONS:
Drug: Sunitinib — Sunitinib: 50mg once daily orally for 4 weeks followed by 2 weeks off treatment (either at 8 a.m. or at 8 p.m.)
  Other Names: Background therapy
Drug: Isoquercetin — Isoquercetin: 225mg twice a day(at 08 a.m. and at 4 p.m)/Isoquercetin: 450 mg twice a day(at 08 a.m. and at 4 p.m).
  Other Names: PR1
  Arms: Experimental Arm
Drug: Placebo — Placebo: 225mg twice a day(at 08 a.m. and at 4 p.m)/Placebo: 450 mg twice a day(at 08 a.m. and at 4 p.m).
  Other Names: PL1
  Arms: Placebo Arm

SUMMARY:
Advanced renal cell carcinoma is invariably fatal, with a life expectancy of 2-3 years since diagnosis. Sunitinib is the standard first-line treatment for this condition, but it is associated to multiple side effects, with fatigue being reported in 51-63% of patients. As sunitinib-induced fatigue is likely to be mediated by inhibition of AMPk function, the investigators hypothesize that isoquercetin, which is hydrolyzed in vivo to quercetin, a known AMPk activator, is able to reduce fatigue in kidney cancer patients taking sunitinib.

DETAILED DESCRIPTION:
Sunitinib is an oral receptor tyrosine kinase inhibitor (TKI) that inhibits vascular endothelial growth factor receptors (VEGFRs), platelet derived growth factor receptor (PDGFRs) and c-kit. Sunitinib was the first TKI to be approved for the first-line treatment of advanced kidney cancer on the grounds of the results achieved in the phase III trial of sunitinib vs. interferon by Motzer et al. in 2007. In this trial, the improvement in quality of life was modest if compared to the advantage in PFS and response rate, which can be related to the multiple adverse events of sunitinib. Sunitinib-induced toxicity includes fatigue, hypertension, bone marrow toxicity, skin toxicity, and gastrointestinal toxicity. Prevalence of fatigue has been reported to be 92% during administration of chemotherapy agents, while in the case of kidney cancer patients treated with sunitinib, fatigue of any grade has been reported in up to 51-63% of patients, with approximately 7% of them showing grade 3-4 fatigue. According to the definition of NCCN guidelines, cancer-related fatigue is a distressing, persistent, subjective sense of physical, emotional, and/or cognitive tiredness or exhaustion related to cancer or cancer treatment that is not proportional to recent activity and interferes with usual functioning. There are a number of general suggestions and behavioral recommendations (e.g. moderate physical activity) that can be easily and effectively implemented in the standard care for treatment and prevention of fatigue in cancer patients. Awareness of these recommendations is still insufficient among physicians. The use of alternative strategies, which include cognitive-behavioral therapies and pharmacological agents may be effective, but present a number of barriers (access to health care workers with appropriate expertise, reimbursement policy, patient's attitude, drug adverse events) that limit their impact in routine clinical practice. The molecular mechanisms of sunitinib-related fatigue are related to off target inhibition of multiple kinases involved in cellular metabolism. In particular, sunitinib inhibits the AMPK enzyme with an IC50 which is in the nanomolar range, thus interfering with catabolic, energy-producing processes, such as glycolysis and lipid oxidation at a systemic level. Furthermore, sunitinib also inhibits GLUT 4-mediated intracellular transport of glucose. For these reasons, sunitinib is likely to cause fatigue via mechanisms which are different with respect to those associated to the underlying cancer and conventional chemotherapy agents. Of note, no randomized, interventional trial has ever been conducted to tackle fatigue in kidney cancer patients treated with sunitinib. The current management of fatigue in these patients remains unsatisfactory at the present time. Quercetin is a naturally occurring flavonol characterized by a phenyl benzo(y)pyrone-derived structure, which belongs to the broader group of polyphenolic flavonoid substances. While quercetin is an aglycone, naturally occurring quercetin compounds are primarily glycosides, with only very small quantity occurring as an aglycone. In particular, isoquercetin is the 3-O- of quercetin. Isoquercetin is hydrolyzed in vivo to form quercetin, which is the reason why the biological effects of quercetin and isoquercetin are pharmacodynamically identical, although isoquercetin is comparatively much more bioavailable than quercetin. Quercetin and isoquercetin are FDA-registered nutritional dietary ingredients suitable for consumption by the general population up to 2 g and 600 mg a day, respectively. For the research purposes of this study, it is noteworthy that quercetin stimulates AMPK in vitro, and it increases GLUT 4 translocation to the cytoplasmic membrane at micromolar concentrations comparable to those possibly achievable with oral administration. These biological effects could positively impact sunitinib-induced fatigue. Quercetin was able to reduce chemotherapy-induced fatigue in mice, while in healthy humans, a randomized, placebo-controlled study showed that supplementation of 500 mg of quercetin twice daily for 7 days provided a statistically significant 13.2% increase in bike-ride time to fatigue.

In conclusion, the following bullet points summarize the background and rationale of this study:

1. sunitinib is the main and most widely used first-line treatment for metastatic kidney cancer and causes fatigue in approximately 50-60% of cases;
2. sunitinib-induced fatigue is likely to be mediated by GLUT-4 and AMPK downregulation;
3. fatigue has a negative impact on quality of life, it increases treatment-related morbidity, it is responsible for treatment delay and interruption, dose reduction and may ultimately reduce sunitinib efficacy;
4. Quercetin is a natural flavonol normally present in food and has been FDA-registered as a nutritional dietary ingredient for the general population up to 1 g per day. Isoquercetin is a quercetin derivative hydrolyzed in vivo to quercetin, and has been considered safe for the general population as a nutritional supplement at a dose of up to 600 mg a day by the FDA. The Institutional Review Board at the Dana-Farber Institution and the FDA have recently approved experimentation of two dose levels of isoquercetin, 500 mg and 1000 mg, to be simultaneously tested in the phase IIb part of a large phase II/III trial for thrombosis prevention in cancer patients (ClinicalTrials.gov: NCT02195232);
5. no significant negative pharmacokinetic /pharmacodynamic interaction during the treatment is expected, as in vivo studies did not show any relevant pharmacokinetic interaction of quercetin with CYP-metabolized drugs;
6. The doses employed in this study are well below the maximum tolerated dose found in a phase I study testing intravenous quercetin (MTD: 1400 mg/m2). In this study, renal toxicity was the main dose limiting toxicity;
7. isoquercetin may reduce fatigue in kidney cancer patients receiving sunitinib on the basis of a molecular rationale, pre-clinical experimental models and clinical data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received no prior systemic therapy other than sunitinib (including interleukin-2, interferon-α, chemotherapy, bevacizumab, mTOR inhibitor sorafenib or other VEGF TKI) for advanced or metastatic RCC. Patients who received adjuvant treatment with a cancer vaccine are eligible.
2. Patients with locally advanced (defined as disease not amenable to curative surgery or radiation therapy) or metastatic renal cell carcinoma of any histology (equivalent to Stage IV RCC according to AJCC staging) for whom treatment with sunitinib is either planned or ongoing. Patients with non-measurable disease are allowed if metastatic disease can be confirmed;
3. Patients for whom treatment with sunitinib is planned must have had a whole body CT scan within 30 days prior to enrollment; patients who are already being treated with sunitinib at the time of enrollment must have had a whole body CT scan showing non progressive disease according to the RECIST criteria within 30 days of enrollment;
4. ECOG PS of 0 or 1;
5. Age ≥18 years;
6. A female is eligible to enter and participate in this study if she is non-childbearing potential or agrees to use adequate contraception;
7. Adequate organ system functions;
8. Total serum calcium concentration <12.0mg/dL;
9. Left ventricular ejection fraction (LVEF) ≥ lower limit of institutional normal (LLN) as assessed by echocardiography (ECHO) or multigated acquisition (MUGA) scan. The same modality used at baseline must be applied for subsequent evaluations;
10. Patient is able to swallow and retain oral tablets;
11. Written informed consent obtained before any screening procedure and according to local guidelines.

Exclusion Criteria:

1. History of another malignancy;
2. History or clinical evidence of central nervous system (CNS) metastases
3. Any clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding or affect absorption of investigational product
4. Unable to tolerate continuous daily administration of 50 mg sunitinib
5. Presence of uncontrolled infection;
6. Serum potassium < lower normal limits;
7. Corrected QT interval (QTc) >480 ms using Bazett's formula;
8. History of cardiovascular conditions within the past 6 months:
9. Poorly controlled hypertension (defined as systolic blood pressure (SBP) of > 150mmHg or diastolic blood pressure (DBP) of > 90mmHg) at baseline
10. History of cerebrovascular accident (CVA) including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months;
11. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
12. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels;
13. Evidence of active bleeding or bleeding diathesis;
14. Significant hemoptysis within 6 weeks prior to first dose of study drug;
15. Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with patient's safety, obtaining informed consent or compliance to the study;
16. Use any prohibited medications within 14 days of the first dose of study medication;
17. Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug;
18. Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of study treatment;
19. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to or sunitinib;
20. Pregnant or lactating female patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug;
21. Clinically significant depression (PHQ-9 score >15), anxiety (GAD score >10), clinically significant insomnia (positivity of ISQ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of activity of isoquercetin as an anti-fatigue agent (FACT-F questionnaire) | At baseline, and at day 70
  To evaluate the activity of isoquercetin as an anti-fatigue agent in patients with kidney cancer receiving sunitinib by using the FACT-F questionnaire after 2 sunitinib cycles.
The maximum tolerated dose of isoquercetin administered concomitantly with sunitinib | From baseline to Day 70
  • The maximum tolerated dose (450/900 mg daily) of isoquercetin administered concomitantly with sunitinib is the primary end point of the phase I part of the trial;

SECONDARY OUTCOMES:
Effect of isoquercetin on quality of life (FACT-G score) | Up to 12 months
  To evaluate the effect of isoquercetin on quality of life as assessed by the FACT-G score
Effect of isoquercetin on serum markers of inflammation (C reactive protein, IL-6, IL10) | Up to 12 months
  To evaluate the effect of isoquercetin on serum markers of inflammation (C reactive protein, IL-6, IL10)
Effect of isoquercetin on dose density and patient compliance, as determined by dose reductions of sunitinib and requirements of schedule modification | Up to 12 months
  To evaluate the effect of isoquercetin on dose density and patient compliance
Safety and tolerability: To evaluate the safety and tolerability (including AEs, SAEs, withdrawal of treatment due to AE, vital signs, ECG and clinical laboratory) | Up to 12 months
Effect of isoquercetin on muscle index (CT scans) | Up to 12 months
  To evaluate the effect of isoquercetin on muscle index using CT scans
Incidence of deep venous thrombosis (doppler ultrasound) | Up to 12 months
  Incidence of deep venous thrombosis, as assessed by doppler ultrasound
Effect of isoquercetin on patient compliance (questionnaire) | Up to 12 months
  To evaluate the effect of isoquercetin on patient compliance will be used a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Di Lorenzo, MD, Principal Investigator
Locations (5):
- Italy (5):
  - Azienda Ospedaliera Cardarelli Divisione Di Oncologia, Napoli, Napoli
  - Ospedale Oncologico Regionale - Centro di Riferimento Oncologico di Basilicata U.O. di Oncologia Medica, Rionero in Vulture, Potenza
  - Fondazione G. Pascale, Naples
  - University Federico II of Naples, Naples
  - Azienda Ospedaliera Ruggi Aragona, Salerno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aparicio LM, Pulido EG, Gallego GA. Sunitinib-induced asthenia: from molecular basis to clinical relief. Cancer Biol Ther. 2011 Nov 1;12(9):765-71. doi: 10.4161/cbt.12.9.18138. PMID 22045104
- [Result] Di Lorenzo G, Porta C, Bellmunt J, Sternberg C, Kirkali Z, Staehler M, Joniau S, Montorsi F, Buonerba C. Toxicities of targeted therapy and their management in kidney cancer. Eur Urol. 2011 Apr;59(4):526-40. doi: 10.1016/j.eururo.2011.01.002. Epub 2011 Jan 14. PMID 21277078
- [Result] Russo GL, Russo M, Ungaro P. AMP-activated protein kinase: a target for old drugs against diabetes and cancer. Biochem Pharmacol. 2013 Aug 1;86(3):339-50. doi: 10.1016/j.bcp.2013.05.023. Epub 2013 Jun 6. PMID 23747347